CLINICAL TRIAL: NCT02835131
Title: Compassionate Use of SOM230 for Individual Patient (NS, 14-Jan-1986) With Hyperinsulinemic/Hypoglycemia
Brief Title: Compassionate Use of SOM230 for Hyperinsulinemic/Hypoglycemia
Status: No longer available | Type: Expanded Access
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Vafa Tabatabaie, Asst Prof. Department of Medicine (Endocrinology), Montefiore Medical Center
Other Study IDs: 2015-5564
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Congenital Hyperinsulinism
Keywords: hyperinsulinemia; hypoglycemia; somatostatin; pasireotide; congenital
MeSH Terms: conditions — Congenital Hyperinsulinism; Hyperinsulinism; Hypoglycemia | interventions — pasireotide

INTERVENTIONS:
Drug: Pasireotide
  Other Names: Signifor; SOM230

SUMMARY:
Congenital hyperinsulinism is a rare condition that can cause life-threatening hypoglycemia. Current treatment for congenital hyperinsulinism is often suboptimal, and such individuals may respond to a new somatostatin analog, pasireotide. This is a compassionate use study of the effects of pasireotide on individuals with suboptimally treated congenital hyperinsulinism.

DETAILED DESCRIPTION:
Congenital hyperinsulinism is a rare condition that can cause life-threatening hypoglycemia. Current treatment for congenital hyperinsulinism is often suboptimal, with diazoxide as the mainstay of treatment. Individuals who are not adequately treated with diazoxide may undergo pancreatectomy. Octreotide has been used with some success in congenital hyperinsulinism but there is limited data on pasireotide, the newest somatostatin receptor agonist, which, compared to octreotide, has 30-40 times greater affinity for somatostatin receptors 1 (SSTR1) and 5 (SSTR5), 5 times greater for somatostatin receptor 3 (SSTR3) and a comparable affinity for somatostatin receptor 2 (SSTR2).

In human islets, SSTR2 & SSTR5 are present in beta cells. Therefore, there is reason to believe that pasireotide may have greater effectiveness than octreotide in preventing hypoglycemia due to hyperinsulinism. Indeed hyperglycemia is a known effect of pasireotide when used for treatment of Cushing's disease and Acromegaly. The current study is of compassionate use for prevention of hypoglycemia in individuals with congenital hyperinsulinemic hypoglycemia who are not adequately treated with diazoxide.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older
2. Patients with a confirmed diagnosis of hyperinsulinemic hypoglycemia, if possible by genetic testing
3. Patients not controlled by medical therapies (e.g. diazoxide or octreotide) and/or pancreatic surgery or patients not eligible for surgery
4. World Health Organization/ Eastern Cooperative Oncology Group Performance Status of 0-2.
5. Life expectancy ≥12 weeks
6. Adequate end organ function as defined by:

   No evidence of significant liver disease:
   * Serum total bilirubin ≤1.5 x upper limit of normal (ULN)
   * International Normalized Ratio (INR) < 1.3
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 2 x ULN,
   * Alkaline phosphatase ≤ 2.5 x ULN
7. Written informed consent obtained prior to treatment to be consistent with local regulatory requirements
8. Is suffering from a serious or life-threatening disease or condition
9. Does not have access to a comparable or satisfactory alternative treatment (i.e., comparable or satisfactory treatment is not available or does not exist)
10. Is not eligible for participation in any of the investigators ongoing clinical trials or has recently completed a clinical trial that has been terminated and, after considering other options (for example., trial extensions, amendments, etc.), the clinical team has determined that treatment is necessary and there are no other feasible alternatives for the patient
11. There are meaningful human clinical data to support an assessment that the potential benefits to patient outweigh risks.
12. Meets any other relevant medical criteria for compassionate use of the investigational product
13. Is not being transferred from an ongoing clinical trial for which they are still eligible

Exclusion Criteria:

1. Patients with a known hypersensitivity to somatostatin analogs or any component of the pasireotide long acting release (LAR) or subcutaneous. formulations.
2. Patients with abnormal coagulation (prothrombin time or activated partial thromboplastin time elevated by 30% above normal limits).
3. Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion.
4. Patients currently using warfarin / warfarin derivatives
5. Patients with symptomatic cholelithiasis.
6. Patients who are not biochemically euthyroid. Patients with known history of hypothyroidism are eligible if they are on adequate and stable replacement thyroid hormone therapy for at least 3 months.
7. QT-related exclusion criteria: :

   * corrected QT interval (QTcF) at screening > 450 msec in males and QTcF > 460 msec
   * History of syncope or family history of idiopathic sudden death
   * Sustained or clinically significant cardiac arrhythmias
   * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular block
   * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), human immunodeficiency virus (HIV) infection, cirrhosis, uncontrolled hypothyroidism or cardiac failure
   * Family history of long QT syndrome
   * Concomitant medications known to prolong the QT interval.
   * Potassium < or = 3.5 mmol/L
8. Patients who have any severe and/or uncontrolled medical conditions :

   * Uncontrolled diabetes as defined by hemoglobinA1c > 8%,
   * Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required; however, previous medical history will be reviewed.
   * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment.
   * Life-threatening autoimmune and ischemic disorders.
9. Patients who have a history of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. Patients who have had no evidence of disease from another primary cancer for 1 or more years are allowed to participate in the study.
10. Patients with history of liver disease, such as cirrhosis or chronic active hepatitis B or
11. Presence of Hepatitis B surface antigen (HbsAg)
12. Presence of Hepatitis C antibody (anti-HCV)
13. History of, or current alcohol misuse/abuse within the past 12 months.
14. Known gallbladder or bile duct disease, acute or chronic pancreatitis
15. Patients with hypomagnesaemia (< 0.7 mmol/L)
16. Patients with a history of non-compliance to medical regimens or who are considered potentially
17. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Combination of any two of the following (a+b or a+c, or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
18. If the patient is a sexually active male he is excluded unless he agrees to use a condom during intercourse while taking pasireotide and for 3 months after stopping pasireotide medication . They should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Vafa Tabatabaie, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States